CLINICAL TRIAL: NCT05795322
Title: Acute Effect of Sound Healing on Pain, Fatigue and Mood: A Retrospective Community Based Study
Brief Title: Acute Effect of Sound Healing on Pain, Fatigue and Mood
Status: Completed | Type: Observational
Sponsor: Innowage Limited (Industry)
Collaborators: Aarogyam UK (Other); Suara Sound Academy (Unknown)
Responsible Party: Sponsor
Other Study IDs: Inn-AA-SS-002
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Pain; Fatigue; Mood Change
Keywords: Sound healing with tuning forks
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tuning for Health: Community based group 'Tuning for Health' was set up to provide chronic condition self-management support to people. Trained, experienced therapist-led group used half an hour of sound healing in virtual session.
  Interventions: Other: Sound healing with tuning forks

INTERVENTIONS:
Other: Sound healing with tuning forks — Over the course of a half-hour virtual session, a specially developed "triple OM track" created by tuning forks was played.

SUMMARY:
There is evidence that sound healing improves health and well-being. However, sound healing modalities, such as tuning forks, continue to be understudied, especially among people with chronic illnesses. This study examined responses to a single session of sound healing and explored whether responses varied based on analogue pain, fatigue, and mood.

ELIGIBILITY:
Inclusion Criteria:

* People with long term illnesses who attended 'Tuning for Health' virtual session

Exclusion Criteria:

* Who did not complete 30-mins Sound Healing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged between 18-85, having long term illnesses for more than 6-month, completed 30-mins selected sound healing track with tuning forks virtually and shared their impact post session, were evaluated retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | From baseline to 30-minutes post intervention
  Visual Analogical Scale (VAS) from 0 to 10 scores where 0 describes no pain and 10 worst pain.
Change in Fatigue | From baseline to 30-minutes post intervention
  Visual Analogue Scale for Fatigue (VAS-F) with18 items relating to the subjective experience of fatigue, with each item representing how they currently feel along a visual analogue scale extending between two extremes (e.g., "not at all tired" to "extremely tired").
Change in Mood | From baseline to 30-minutes post intervention
  Visual Analogue Mood Scale using vertical 100 mm lines and schematic faces representing the following mood states: sad, afraid, angry, tired, energetic, happy, and confused.

SECONDARY OUTCOMES:
Patients Satisfaction | From baseline to 30-minutes post intervention
  Patients Satisfaction was measured using 5-Linkert Scale (Very dissatisfied, Somewhat dissatisfied, Neutral, Somewhat satisfied, Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Debbi Walker, Study Director — Suara Sound Academy; Neha Sharma, PhD, Principal Investigator — Aarogyam UK CIC
Locations (1):
- Aarogyam UK CIC, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided